CLINICAL TRIAL: NCT04214457
Title: Prospective, National and Multicenter Biomedical Study of Cohorts, Aimed at Patients With Surgical Indication of Hysterectomy, Laparoscopic or Laparotomic Myomectomy Due to Diagnosis of Myometrial Tumors (Leiomyoma / Leiomyosarcoma)
Brief Title: Development of a Predictive Model for Early Differential Diagnosis of Uterine Leiomyomas and Leiomyosarcomas
Acronym: MYOSARC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX1-MYO-CS-19-03
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Leiomyoma; Leiomyosarcoma
Keywords: Leiomyoma (LM); Leiomyosarcoma (LMS); Next Generation Sequencing (NGS); Circulating tumor DNA (ctDNA)
MeSH Terms: conditions — Leiomyoma; Leiomyosarcoma | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myometrial tumor with suspected leiomyosarcoma: Women between 18 and 75 years of age diagnosed with a myometrial tumor (probably leiomyoma) with suspected leiomyosarcoma
  Interventions: Procedure: Biopsy and peripheral blood collection

INTERVENTIONS:
Procedure: Biopsy and peripheral blood collection — After obtaining informed consent, the samples (tumor tissue and peripheral blood) will be collected at the time of surgery, which the patient had already planned by medical indication according to the usual clinical practice. Part of the sample will be sent to histopathology for gold standard diagnosis while the rest of the sample will be sent to Igenomix for molecular analysis.
  If samples are available from patients who underwent surgery prior to the study, after they sign the Informed Consent, the samples will be sent to Igenomix for molecular analysis and the results obtained by histopathology will be collected from the patient's medical record.

SUMMARY:
The development of an accurate and non-invasive diagnostic method is a priority in areas such as gynecology and oncology, specifically to improve the health of those patients with surgical indication for diagnosis of myometrial tumors: leiomyomas and/or leiomyosarcomas.

Recently, Next Generation Sequencing (NGS) technology has been successfully applied in different areas of knowledge, being effective not only for the detection of DNA mutations, but also providing through bioinformatic tools, new insights in the understanding of chromosomal instability. In addition, the detection of circulating tumor DNA (ctDNA) through this type of techniques could revolutionize the non-invasive detection and monitoring of this type of tumors.

The proposed study aims to perform the differential molecular analysis of myometrial tumor tissue (uterine leiomyomas / leiomyosarcomas), as well as peripheral blood of a group of patients with surgical indication of hysterectomy, laparoscopic or laparotomic myomectomy by diagnosis of myometrial tumors. Thus, the obtained samples will be processed for the realization of techniques of massive parallel sequencing or NGS that, together with a specialized bioinformatic software, will facilitate the interpretation of the obtained data.

Combination of both platforms, sequencing and bioinformatics, will offer a high potential for the discovery of genetic variants and genomic markers. Depending on the results of these analyses, differential diagnosis of leiomyoma and leiomyosarcoma could be determined, in addition to increasing knowledge of myometrial biology and associated pathologies in a clinical and therapeutic context. Moreover, the application of this technology could allow the development of biomarkers and targeted therapies effective in the treatment of uterine leiomyomas and/or leiomyosarcomas.

DETAILED DESCRIPTION:
Leiomyomas (LM) are the most common benign gynecological tumors that affect approximately 70% of women of reproductive age, being responsible for 200,000 hysterectomies per year in the United States (USA). Despite its benign nature, LM represents a major public health problem due to its significant level of morbidity, which manifests as a spectrum of clinical symptoms such as heavy menstrual bleeding, anemia, pelvic pain, infertility and recurrent pregnancy loss, among others.

Uterine leiomyosarcoma (LMS) is a rare uterine malignancy that arises from the smooth muscle of uterine wall. It accounts for only 1-2% of uterine malignancies and occurs mainly after menopause. LMS is notorious for its aggressive nature and poor prognosis.

Although uterine LM and LMS are considered biologically unrelated tumors due to their cytogenetic and molecular disparity, both share morphological features that can complicate the diagnosis through current clinical tests or factors.

Nowadays, long-term therapeutic options for LM are limited. Currently, laparoscopic morcellation is the most widely used surgical technique in the treatment of large LM. However, this type of surgery carries the risk of occult dissemination of malignant tumors such as LMS, characterized by early metastases, poor prognosis and high recurrence rates, with limited therapeutic efficacy. In fact, the United States Food and Drug Administration (FDA) has estimated that 1 in 352 of women with surgical indication of LM could have LMS, and treatment in this case could result in tumor spread. Given this need, Igenomix, through a recent pilot study with 26 samples, has identified new genetic targets that potentially differentiate leiomyosarcomas and leiomyomas, through integrated comparative genomic and transcriptomic analyses. This allowed to lay the foundations, not only to improve the understanding of the pathogenesis of these uterine tumors, but also provides a first step towards the preoperative diagnosis of leiomyomas and leiomyosarcomas by liquid biopsy.

Based on this pilot study, a new clinical study is proposed to proceed with further identification of genetic markers and develop a preoperative diagnosis of LM and LMS by liquid biopsy. A total sample size of 1,000 patients with suspected LMS is expected to be recruited in this study, considering the frequency of surgeries in which obtaining a sample is intended, as well as the frequency of patients who will accept tissue donation for research. Moreover, a cut-off point with a preliminary analysis every 100 patients will be established, in which the laboratory data is combined with those derived from the Pathological Anatomy (Gold Standard), so that when a total of 40 LMS is reached the study will end.

During the development of the study, after obtaining informed consent from eligible patients, the samples (tumor tissue and peripheral blood) will be collected at the time of surgery, which the patient had already planned by medical indication according to the usual clinical practice. Thus, the participation of the subject in this study will entail only a single visit coinciding with the day of the surgery. In addition, samples available from patients that underwent surgery before the study could be also included if, after being duly informed, the patient agrees to participate in the study and signs the study consent form. Exceptionally, samples from patients who could not consent due to major reasons (such as death of the subject or impossibility to be found) could also be included in the study upon approval of the appropriated Ethic Committee according to the local regulations for this type of situations. In any case, the investigators will ensure that there is no expressed objection from the donors in their clinical history and that samples will be codified in order to assure anonymity.

Samples will be sent to histopathological diagnosis and to Igenomix, that will develop and optimize laboratory protocols to detect changes at the DNA (Whole Exome Sequencing) and RNA (RNAseq) level in order to achieve the described outcomes. This new approaches focused on NGS, could allow not only the detection of tumor-specific mutations but, in combination with bioinformatics tools, could provide new knowledge to understand chromosomal instability in the tumors.

According to the histopathological diagnosis, patients will be treated by their respective doctors and followed up to determine their evolution. If the proposed hypothesis from NGS results is confirmed and the objectives are achieved, in a second phase of the project, a diagnostic tool will be developed to extend the non-invasive genetic diagnosis of uterine leiomyomas and leiomyosarcomas in peripheral blood through the free DNA analysis of circulating tumor cells. The possibility of being able to quantify and characterize the circulating tumor DNA (ctDNA) by means of this type of techniques, could revolutionize the non-invasive detection and the follow-up of this type of tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily sign the informed consent approved by the research Ethics Committee (EC) after having been duly informed of the nature of the study, before carrying out any test, knowing the potential risks, benefits and discomforts arising from their participation. Participants should be informed that they may leave the study at any time, without this implying any consequences for their subsequent medical care.
* Body Mass Index (BMI) = 18-35 kg/m2
* Age = 18-75 years
* Surgical indication of hysterectomy, laparoscopic or laparotomic myomectomy by imaging diagnosis (ultrasound, resonance, Computerized Tomography Scan ...) of tumor mass in the myometrium, whether primary or recurrent.

Exclusion Criteria:

* Patients who have participated in another biomedical study or who have received an experimental treatment during the last 30 days, unless approved by the sponsor.
* Patients who have received chemotherapy or radiotherapy 6 months before diagnosis (in case of recurrence).
* Pregnant patients before or during the development of the study.
* Existence of serious or uncontrolled bacterial, fungal or viral infections that, in the opinion of the principal investigator, may interfere with the patient's participation in the study or in the evaluation of the study results.
* Any illness or medical condition that is unstable or could endanger the patient's safety and compliance in the study.
* Psychological, family, sociological or geographical situations that do not allow compliance with the protocol or the signing of informed consent.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women between 18 and 75 years of age and BMI between 18-35 kg/m2, diagnosed with a myometrial tumor (probably leiomyoma) with suspected leiomyosarcoma, will be evaluated at their reference center, verifying that they comply the inclusion / exclusion criteria to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Identification of specific genetic markers for leiomyomas and leiomyosarcomas | 36 months
  Identification of genetic markers that allow the classification of myometrial tumors into leiomyomas and leiomyosarcomas by NGS.

SECONDARY OUTCOMES:
Characterization of cell populations of uterine leiomyomas and leiomyosarcomas | 36 months
  Single-cell DNA/RNAseq characterization of the uterine leiomyomas and leiomyosarcomas cell populations in order to assess the heterogeneity in these myometrial tumors.
Identification of methylation patterns characteristic of the tumorigenic process | 36 months
  Study of methylation patterns that could identify tumorigenic processes

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simón, MD, PhD, Study Chair — Igenomix; Aymara Mas, PhD, Principal Investigator — Igenomix Foundation
Locations (4):
- Spain (4):
  - Complejo Hospitalario Universitario de Cartagena, Cartagena, Murcia
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No